CLINICAL TRIAL: NCT05456932
Title: Predicting Response to Iron Supplementation in Patients With Active Inflammatory Bowel Disease
Acronym: PRIme
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: University Medical Center Groningen (Other); Radboud University Medical Center (Other); Maastricht University Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Andrea E. van der Meulen - de Jong, MD, PhD, Principal Investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL79105.058.22; 2022-000894-16 (EudraCT Number)
Record Dates: First submitted 2022-05-10; First posted 2022-07-13 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Inflammatory Bowel Diseases; Iron-deficiency; Iron Deficiency Anemia
Keywords: IBD; Crohn's disease; Ulcerative colitis; Inflammatory Bowel Disease; Iron deficiency; Iron deficiency anemia
MeSH Terms: conditions — Inflammatory Bowel Diseases; Anemia, Iron-Deficiency; Crohn Disease; Colitis, Ulcerative; Iron Deficiencies | interventions — ferric maltol; ferrous fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intravenous iron (Experimental): Intravenous iron therapy
  Interventions: Drug: Intravenous iron
- Ferric maltol (Experimental): Treatment with oral ferric maltol
  Interventions: Drug: Ferric maltol
- Ferrous fumarate (Experimental): Treatment with oral ferrous fumarate
  Interventions: Drug: Ferrous fumarate

INTERVENTIONS:
Drug: Intravenous iron — Included participants will receive intravenous iron therapy, the dosage will be based on national pharmaceutical formulary.
  Other Names: i.v. iron
  Arms: Intravenous iron
Drug: Ferric maltol — Included participants will receive oral iron therapy with ferric maltol (twice a day 30mg for 12 weeks)
  Other Names: Feraccru
  Arms: Ferric maltol
Drug: Ferrous fumarate — Included participants will receive oral iron therapy with ferrous fumarate (twice a day 100mg for 12 weeks)
  Other Names: ferrofumaraat
  Arms: Ferrous fumarate

SUMMARY:
Iron deficiency anemia is the most common systemic manifestation of Inflammatory Bowel Diseases (IBD)-Crohn's disease and ulcerative colitis. Iron deficiency with or without anemia poses a diagnostic and therapeutic challenge due to chronic gastrointestinal blood loss and the inflammatory nature of IBD. Recent illumination of iron metabolism has brought attention to the systemic iron regulator-hepcidin, a peptide hormone that regulates intestinal iron absorption and systemic iron availability. Elevated hepcidin is associated with oral iron malabsorption in IBD. This study aims to evaluate whether hepcidin concentration at baseline can predict response to oral and intravenous iron therapy in patients with IBD and concomitant iron deficiency with or without anemia.

DETAILED DESCRIPTION:
The PRIme is a multicenter and randomized study that aims to evaluate the capacity of hepcidin at baseline to predict response to oral or intravenous iron therapy in patients with active IBD. Study participants will be randomized and allocated (open-label) to one of the three study arms: intravenous iron therapy, therapy with oral ferrous fumarate, or therapy with oral ferric maltol.

During the study, biochemical indices such as hemoglobin, iron status, hepcidin and related cytokines will be measured at week 6, 14, and 24 after the start of the therapy. In addition, the study will evaluate changes in oxidative stress, quality of live, and productivity.

ELIGIBILITY:
Inclusion Criteria:

* Established IBD diagnosis (Crohn's disease, ulcerative colitis, IBD-unclassified)
* Adults (≥18 years of age)
* Active IBD (defined as any endoscopic, radiologic or biochemical disease activity [fecal calprotectin >150 mg/kg or C-reactive protein >5 mg/l])
* Iron deficiency anemia (defined as ferritin <100 ug/l and hemoglobin <7.5 mmol/l for females or <8.5 mmol/l for males) or iron deficiency (defined as ferritin <100 ug/l and transferrin saturation <20%)
* Documented informed consent

Exclusion Criteria:

* Blood transfusion or therapy with oral and/or intravenous iron in the past eight weeks
* Documented intolerance to oral or intravenous iron
* Severe anemia (defined as hemoglobin <6.2 mmol/l for females and males)
* Documented history of liver cirrhosis, heart failure, hemoglobinopathies, autoimmune hemolytic anemia, myelodysplastic syndrome, or chronic obstructive pulmonary disease
* Documented history of recent treatment for a malignancy (excluding dermatological malignancies such as basal cell carcinoma or squamous cell carcinoma). Patients can be included if the treatment for malignancy has been finalized ≥6 months before the inclusion date.
* Documented history of bariatric surgery or gastric/duodenal resections due to benign or malignant pathologies
* End-stage renal disease (impaired renal function, defined as estimated Glomerular Filtration Rate (eGFR) <30 ml/min/1.73m2)
* Folic acid deficiency
* Vitamin B12 deficiency
* Documented pregnancy or breastfeeding at the time of inclusion
* Documented major operation (e.g., laparotomy) less than six weeks before inclusion
* Unable to give informed consent due to inability to understand Dutch language or incapacitation (e.g., due to cognitive/psychological conditions or hospitalization in Intensive Care)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-08-19 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
The discriminative capacity of hepcidin at baseline to differentiate between response and non-response to iron therapy with oral ferrous fumarate | Week 14
  Hepcidin concentration will be measured in blood at baseline. Receiver Operating Characteristic (ROC) curve with associated Area Under the Curve (AUC) will be used to evaluate the discriminative ability of hepcidin concentration at baseline to differentiate between response and non-response to iron therapy with ferrous fumarate. Response to iron therapy will be evaluated at week 14 and will be defined as hemoglobin normalization (or >1.2 mmol/L increase) for patients with iron-deficiency anemia; for patients with non-anemic iron deficiency the response will be defined as normalization of iron stores (i.e., ferritin >100 ug/L and transferrin saturation >20%).
The discriminative capacity of hepcidin at baseline to differentiate between response and non-response to iron therapy with oral ferric maltol | Week 14
  Hepcidin concentration will be measured in blood at baseline. Receiver Operating Characteristic (ROC) curve with associated Area Under the Curve (AUC) will be used to evaluate the discriminative ability of hepcidin concentration at baseline to differentiate between response and non-response to iron therapy with ferric maltol. Response to iron therapy will be evaluated at week 14 and will be defined as hemoglobin normalization (or >1.2 mmol/L increase) for patients with iron-deficiency anemia; for patients with non-anemic iron deficiency the response will be defined as normalization of iron stores (i.e., ferritin >100 ug/L and transferrin saturation >20%).
The discriminative capacity of hepcidin at baseline to differentiate between response and non-response to intravenous iron therapy | Week 14
  Hepcidin concentration will be measured in blood at baseline. Receiver Operating Characteristic (ROC) curve with associated Area Under the Curve (AUC) will be used to evaluate the discriminative ability of hepcidin concentration at baseline to differentiate between response and non-response to intravenous iron therapy. Response to iron therapy will be evaluated at week 14 and will be defined as hemoglobin normalization (or >1.2 mmol/L increase) for patients with iron-deficiency anemia; for patients with non-anemic iron deficiency the response will be defined as normalization of iron stores (i.e., ferritin >100 ug/L and transferrin saturation >20%).

SECONDARY OUTCOMES:
Change in hepcidin | weeks 6, 14, and 24
  Change in hepcidin levels from baseline to weeks 6, 14, and 24 in all of the three groups
Change in soluble Transferrin Receptor (sTfR) | weeks 6, 14, and 24
  Change in soluble Transferrin Receptor (sTfR) levels from baseline to weeks 6, 14, and 24 in all of the three groups.
Change in interleukin 6 (IL-6) | weeks 6, 14, and 24
  Change in interleukin 6 (IL-6) levels from baseline to weeks 6, 14, and 24 in all of the three groups.
Normalization of iron stores | weeks 6, 14, and 24
  Percentage of patients who achieve normalization of iron stores (an increase in transferrin saturation (transferrin saturation >20%) and an increase in ferritin above 100 ug/l) at weeks 6, 14, and 24 in all of the three groups.
Correlation between response to iron therapy and disease activity | week 14
  The correlation of disease activity (evaluated by fecal calprotectin levels) and response to iron therapy in all of the three groups.
Incidence of hypophosphatemia during iron therapy | weeks 6, 14, and 24
  Percentage of patients who experienced hypophosphatemia throughout iron therapy in all of the three groups
Adverse events during iron therapy | weeks 6, 14, and 24
  Number of (serious) adverse events in all of the three groups.
Change in clinical disease activity | weeks 14 and 24
  Change in clinical disease activity (measured by mobile Health Index (mHI) 0-24 for patients with Crohn's disease and 0-34 for patients with ulcerative colitis; higher scores indicate a more active disease) from baseline to week 14, and week 24 in all of the three groups.
Change in quality of life | weeks 14 and 24
  Change in quality of life (measured by 36-item Short Form Survey (SF-36) expressed on a scale 0-100 where higher scores indicate less disability and better quality of life) from baseline to week 14, and week 24 in all of the three groups.
Change in activity and productivity | weeks 14 and 24
  Change in activity and productivity (measured by Work Productivity and Activity Impairment: Inflammatory Bowel Disease (WPAI:IBD) expressed as 0-100% where higher percentages indicate greater impairment) from baseline to week 14, and week 24 in all of the three groups.
Hematologic response during iron therapy | weeks 14 and 24
  Percentage of patients who achieved an adequate hematologic response (defined by hemoglobin increase >1.2 mmol/L or hemoglobin normalization) at weeks 14 and 24 in all of the three groups.
Hemoglobin increase (>0.6 mmol/L) during iron therapy | weeks 6 and 14
  Percentage of patients who experienced a ≥0.6 mmol/l change in hemoglobin from baseline to weeks 6 and 14 in all of the three groups.

OTHER OUTCOMES:
Exploratory outcome: change in oxidative stress | weeks 6, 14, and 24
  Change in oxidative stress (measured by free-thiol levels) from baseline to week 6, week 14.

CONTACTS AND LOCATIONS:
Overall Officials: A.E. van der Meulen - de Jong, MD, PhD, Principal Investigator — LUMC
Locations (5):
- Netherlands (5):
  - Amsterdam University Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center (LUMC), Leiden
  - Maastricht University Medical Center+, Maastricht
  - Radboud University Medical Center, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Loveikyte R, Duijvestein M, Mujagic Z, Goetgebuer RL, Dijkstra G, van der Meulen-de Jong AE. Predicting response to iron supplementation in patients with active inflammatory bowel disease (PRIme): a randomised trial protocol. BMJ Open. 2024 Jan 30;14(1):e077511. doi: 10.1136/bmjopen-2023-077511. PMID 38296290